CLINICAL TRIAL: NCT00459706
Title: A 3-Month, Randomised, Open-Label, Parallel-Group, Descriptive Study To Explore And Compare Perceptions and Satisfaction For Two Different Delivery Mechanisms For Etanercept (Etanercept Autoinjector And The Etanercept Prefilled Syringe) In Patients With Rheumatoid Arthritis
Brief Title: Study Comparing Perceptions and Satisfaction for Two Different Delivery Mechanisms for Etanercept
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881K1-6000; B1801017 (Other: Pfizer); NCT00595452 (obsolete NCT alias)
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Results first posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

ARMS (2):
- Enbrel 50 mg Prefilled Syringe (Experimental): Enbrel 50 mg subcutaneously once weekly for 12 Weeks using Prefilled Syringe
  Interventions: Device: Enbrel 50 mg Prefilled Syringe
- Enbrel 50 mg Autoinjector (Experimental): Enbrel 50 mg subcutaneously once weekly for 12 Weeks using Autoinjector
  Interventions: Device: Enbrel 50 mg Autoinjector

INTERVENTIONS:
Device: Enbrel 50 mg Prefilled Syringe — Enbrel 50 mg subcutaneously once weekly for 12 Weeks using Prefilled Syringe
  Arms: Enbrel 50 mg Prefilled Syringe
Device: Enbrel 50 mg Autoinjector — Enbrel 50 mg subcutaneously once weekly for 12 Weeks using Autoinjector
  Arms: Enbrel 50 mg Autoinjector

SUMMARY:
The purpose of this study is to explore and compare the perceptions and satisfaction for two different delivery mechanisms for Etanercept (Etanercept Autoinjector and the Etanercept Prefilled Syringe) in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This study describes patient perceptions related to device attributes, which are of importance in describing overall patient perception. A range of potential device benefits (e.g. ease of use, convenience, confidence, presence or absence of fear, side effects related to administration) is captured using a questionnaire based on the outputs of patient interviews.

The study aims to characterize patient attributes that will indicate when one device may result in greater patient satisfaction than another. Patient attributes are composed of patient characteristics (e.g. age, sex, self efficacy, expectations of treatment, perception of their illness) and RA characteristics (e.g. disease severity, disease duration, prior treatment, functional impairment).

ELIGIBILITY:
Inclusion:

* Diagnosis of RA according to the ACR-Criteria.
* Eligible for treatment with etanercept according to Summary of Product Characteristics (SmPC), and applicable local guidelines.
* Willing and able to self-inject etanercept.

Exclusion:

* Prior experience of biologics and anti-TNF treatment for their RA including etanercept.
* Sepsis or risk of sepsis.
* Current or recent infections, including chronic or localized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (106):
- Denmark (4):
  - Frederiksberg
  - Hjørring
  - Holbæk
  - Silkeborg
- Finland (4):
  - Helsinki
  - Hyvinkää
  - Joensuu
  - Lohja
- France (20):
  - Amiens
  - Aulnay-sous-Bois
  - Avignon
  - Boulogne-Billancourt
  - Brest
  - Cahors
  - Corbeilles-Essonnes
  - Grenoble
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Niort
  - Orléans
  - Paris
  - Pierre-Bénite
  - Reims
  - Rouen
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (22):
  - Erlangen, Bay
  - Frankfurt am Main, Hesse
  - Pirna, Saxony
  - Bad Abbach
  - Bad Nauheim
  - Berlin
  - Cologne
  - Düsseldorf
  - Erlangen
  - Essen
  - Göttingen
  - Hanover
  - Hofheim/Taunus
  - Leipzig
  - München
  - Nienburg
  - Oberammergau
  - Osnabrück
  - Tübingen
  - Villingen-Schwenningen
  - Würzburg
  - Zeven
- Italy (27):
  - Ariano Irpino, Avellino
  - S. Pietro Vernotico, Brescia
  - San Cesario di Lecce, Lecce
  - Alessandria
  - Bologna
  - Cagliari
  - Cinisello Balsamo
  - Como
  - Coppito
  - Fano
  - Ferrara
  - Foggia
  - Massa
  - Milan
  - Napoli
  - Padua
  - Palermo
  - Parma
  - Reggio Calabria
  - Rieti
  - Roma
  - S. Dona Di Piave
  - Terni
  - Torino
  - Torrette Di Ancona
  - Verona
  - Vimercate
- Netherlands (3):
  - Arnhem
  - Eindhoven
  - Rotterdam
- Norway (7):
  - Gjettum
  - Harstad
  - Kristiansand
  - Lillehammer
  - Skien
  - Trondheim
  - Tønsberg
- Sweden (7):
  - Danderyd
  - Malmo
  - Stockholm
  - Sundsvall
  - Uppsala
  - Vasterås
  - Västerås
- United Kingdom (12):
  - Ashford
  - Basingstoke
  - Cambridge
  - Chertsey
  - London
  - Manchester
  - Portsmouth
  - Southampton
  - Stoke-on-Trent
  - Truro
  - Westcliff-on-Sea
  - Wigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Enbrel 50 mg Autoinjector: Enbrel 50 milligram (mg) once weekly subcutaneously for 12 Weeks using autoinjector
- Enbrel 50 mg Prefilled Syringe: Enbrel 50 mg once weekly subcutaneously for 12 Weeks using prefilled syringe
Period: Overall Study
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Started | 325 | 315
MODIFIED INTENT-TO-TREAT POPULATION | 324 (1 participant had no evaluation after the first injection) | 313 (2 participants withdrew consent before the first injection)
Completed | 299 | 294
Not Completed | 26 | 21
Not completed — Adverse Event | 19 | 13
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Physician Decision | 2 | 0
Not completed — Discontinuation of Study by Sponsor | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Failed to Return | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Enbrel 50 mg Autoinjector: Enbrel 50 mg once weekly subcutaneously for 12 Weeks using autoinjector
- Total: Total of all reporting groups
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe | Total
Number analyzed (Participants) | 325 | 315 | 640
Age Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.9) | 54.8 (12.9) | 54.7 (12.9)
Sex/Gender, Customized [Number; unit: participants]
  Male | 85 | 78 | 163
  Female | 240 | 237 | 477

OUTCOME MEASURES:

1. Primary Outcome: Participant Satisfaction on Day 84 for 2 Different Delivery Mechanisms for Etanercept, Modified Intent-to-treat Population
Description: Participant's response to the question "How satisfied are you with your injection device?" scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher score indicated greater satisfaction with the delivery mechanism.
Time Frame: Day 84
Population: Modified Intent-to-Treat (mITT): All randomized participants who received at least 1 injection of test article and had at least 1 available evaluation after the first administration of test article. Number of participants analyzed (N) = participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 306 | 300
units on a scale | 8.3 (2.4) | 7.2 (2.6)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Non-inferiority of autoinjector (AI) over prefilled syringe (PFS) was assessed on the primary endpoint. Hypothesis tested was H0: AI minus PFS less than or equal to (≤) -1. The alternate hypothesis was H1: AI minus PFS greater than (>) -1; Test type: Non-Inferiority or Equivalence — The non-inferiority test was performed using the 95 percent (%) two-sided confidence interval (CI) of the difference (AI minus PFS) of mean subject satisfactions (α = 2.5%). Non-inferiority was demonstrated if the lower limit of the two-sided 95% CI > -1; p < 0.001, ANOVA; ANOVA=analysis of variance; Mean Difference (Net) = 1.11, 95% CI 2-sided [0.71 to 1.50], Standard Error of Mean 0.20

2. Primary Outcome: Participant Satisfaction on Day 84 for 2 Different Delivery Mechanisms for Etanercept, Per-Protocol Population
Description: as for outcome 1
Time Frame: Day 84
Population: Per-protocol (PP): mITT participants who completed the study with no major protocol violation. N=participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 292 | 281
units on a scale | 8.4 (2.2) | 7.2 (2.6)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Non-inferiority of AI over PFS was assessed on the primary endpoint. The hypotheses tested was as follows: H0: AI - PFS ≤ -1 H1: AI - PFS > -1; Test type: Non-Inferiority or Equivalence — The non-inferiority test was performed using the 95% two-sided CI of the difference (AI minus PFS) of mean subject satisfactions (α = 2.5%). Non-inferiority was demonstrated if the lower limit of the two-sided 95% CI > -1; p < 0.001, ANOVA; Mean Difference (Net) = 1.25, 95% CI 2-sided [0.85 to 1.64], Standard Error of Mean 0.20

3. Secondary Outcome: Percentage of Participants on Day 28 Satisfied With Either of the Different Delivery Mechanisms for Etanercept
Description: Percentage of participants answering "Yes" to the question "Are you satisfied with your injection device?"
Time Frame: Day 28
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 297
percentage of participants | 92.7 | 88.6
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.058, GEE Model+Logit Link+Binomial Distributn; GEE=Generalized estimating equation Distribn=distribution; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.98 to 3.05]

4. Secondary Outcome: Percentage of Participants on Day 84 Satisfied With Either of the Delivery Mechanisms for Etanercept
Description: Percentage of participants answering "Yes" to the question "Are you satisfied with your injection device?"
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 297 | 284
percentage of participants | 93.3 | 87.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.019, GEE Model+Logit Link+Binomial Distributn; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.12 to 3.43]

5. Secondary Outcome: Participant Satisfaction by Age for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. Results are reported by age categories: <=46 years, >46-55 years, >55-65 years, >65 years.
Time Frame: Day 84
Population: mITT; last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  <=46 years | 8.18 (2.52) | 6.58 (2.73)
  >46 - 55 years | 8.81 (1.84) | 7.01 (2.70)
  >55 - 65 years | 8.31 (2.44) | 7.56 (2.57)
  >65 years | 7.74 (2.54) | 7.63 (2.28)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.160, Regression, Linear; Regression coefficient = 0.11, 95% CI 2-sided [-0.04 to 0.27]

6. Secondary Outcome: Participant Satisfaction by Gender for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism.
Time Frame: Day 84
Population: mITT; LOCF. N=total evaluable participants. n=participants evaluable in that category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  Male (n=85, 77) | 8.45 (2.31) | 8.13 (2.07)
  Female (n=239, 236) | 8.21 (2.40) | 6.89 (2.72)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Female versus male (reference); Test type: Superiority or Other; p = 0.001, Regression, Linear; Regression coefficients = -0.75, 95% CI 2-sided [-1.20 to -0.29]

7. Secondary Outcome: Participant Satisfaction by Socio-Educational Level for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. Participants were categorized into those having only reading/writing capacity, those at the high-school/baccalaureate level, and those at the university level.
Time Frame: Day 84
Population: mITT; LOCF. N=total participants with evaluable data. n=participants with evaluable data for that category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 323 | 311
units on a scale
  Only Reading/Writing Capacity (n=122, 129) | 8.11 (2.24) | 7.53 (2.44)
  High School/Baccalaureate Level (n=147, 136) | 8.32 (2.50) | 6.90 (2.87)
  University Level (n=54, 46) | 8.44 (2.36) | 7.09 (2.38)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Participants at High School/Baccalaureate Level versus participants with only Reading/Writing Capacity (reference); Test type: Superiority or Other; p = 0.676, Regression, Linear; Regression coefficient = -0.18, 95% CI 2-sided [-0.62 to 0.26]
Statistical Analysis 2: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Participants at University Level versus participants with only Reading/Writing Capacity (reference); Test type: Superiority or Other; p = 0.676, Regression, Linear; Regression coefficient = 0.00, 95% CI 2-sided [-0.59 to 0.60]

8. Secondary Outcome: Participant Satisfaction by the Hospital Anxiety Depression (HAD) Anxiety Subscale Score for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. The HAD scale assessed participants' levels of anxiety and depression over the past week; total 14 questions, odd-numbered questions related to anxiety. Responses scored on a 4-point scale; each question was graded in a different way. Anxiety subscale scores ranged from 0 to 21. Lower HAD Anxiety subscale scores indicated better health. Categories are anxiety subscale scores.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  HAD anxiety subscale score <=4 | 8.56 (2.29) | 7.67 (2.44)
  HAD anxiety subscale score >4 - 7 | 8.13 (2.47) | 7.32 (2.56)
  HAD anxiety subscale score >7 - 10 | 7.87 (2.68) | 6.93 (2.53)
  HAD anxiety subscale score >10 | 8.46 (2.06) | 6.67 (2.97)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.020, Regression, Linear; Regression coefficient = -0.28, 95% CI 2-sided [-0.52 to -0.05]

9. Secondary Outcome: Participant Satisfaction by the HAD Depression Subscale Score for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. The HAD scale assessed participants' levels of anxiety and depression over the past week; total 14 questions, even-numbered questions related to depression. Responses scored on a 4-point scale; each question was graded in a different way. Depression subscale scores ranged from 0 to 21. Lower HAD Depression subscale scores indicated better health. Categories are depression subscale scores.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  HAD depression subscale score <=3 | 8.75 (2.02) | 7.70 (2.37)
  HAD depression subscale score >3 - 5 | 7.97 (2.58) | 7.35 (2.66)
  HAD depression subscale score >5 - 8.2 | 8.28 (2.39) | 7.17 (2.49)
  HAD depression subscale score >8.2 | 8.03 (2.48) | 6.23 (2.94)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.008, Regression, Linear; Regression coefficient = -0.35, 95% CI 2-sided [-0.61 to -0.09]

10. Secondary Outcome: Participant Satisfaction by Patient Activation Measure (PAM) Score for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the delivery mechanism. The 13-item short form of the PAM survey assessed participants' knowledge, skill, and confidence for self-management; calibrated scale score ranged from 0 to 100. Higher scores indicated more confidence in managing participants' condition and lifestyle. Results reported by PAM score: <=49.9, >49.9-56.4, >56.4-66, >66.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  PAM scale score <=49.9 | 7.91 (2.58) | 7.06 (2.72)
  PAM scale score >49.9 - 56.4 | 8.48 (2.14) | 7.42 (2.36)
  PAM scale score >56.4 - 66 | 8.02 (2.56) | 6.97 (2.83)
  PAM scale score >66 | 8.49 (2.32) | 7.38 (2.63)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.030, Regression, Linear; Regression coefficient = 0.17, 95% CI 2-sided [0.02 to 0.32]

11. Secondary Outcome: Participant Satisfaction by Prior Self-Injection Experience for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Participants were grouped into 2 categories: those who did and did not have prior self-injection experience. Higher scores indicated greater satisfaction in the delivery mechanism.
Time Frame: Day 84
Population: mITT; LOCF. N=total evaluable participants. n=evaluable participants for that category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  Self-Injection Experience (n=97, 101) | 8.10 (2.51) | 6.57 (2.51)
  No Self-Injection Experience (n=227, 212) | 8.34 (2.32) | 7.49 (2.64)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Self-injection Experience versus No Self-injection Experience (reference); Test type: Superiority or Other; p = 0.006, Regression, Linear; Regression coefficient = -0.60, 95% CI 2-sided [-1.03 to -0.18]

12. Secondary Outcome: Participant Satisfaction by Duration of Rheumatoid Arthritis (RA) for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the delivery mechanism. Results are reported by duration of RA: <=3 years, >3-6 years, >6-13 years, >13 years.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  RA duration <=3 years | 7.99 (2.56) | 7.32 (2.59)
  RA duration >3 - 6 years | 8.39 (2.34) | 6.68 (2.83)
  RA duration >6 - 13 years | 8.52 (2.37) | 7.24 (2.67)
  RA duration >13 years | 8.29 (2.14) | 7.40 (2.47)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.278, Regression, Linear; Regression coefficient = 0.06, 95% CI 2-sided [-0.05 to 0.18]

13. Secondary Outcome: Participant Satisfaction by 28-joint Disease Activity Score (DAS28) for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the delivery mechanism. DAS28 includes a 28 tender joint count, a 28 swollen joint count, erythrocyte sedimentation rate, and a general health assessment on a visual analog scale. Score ranged from 0 to 9.4. Interpretation: disease activity is low when score ≤3.2, moderate when 3.2<score≤5.1, or high when score >5.1, remission when score <2.6. Results are reported by categories of DAS28 score: <=4.7, >4.7-5.4, >5.4-6.2, >6.2.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  DAS28 score <=4.7 | 8.24 (2.50) | 7.01 (2.50)
  DAS28 score >4.7 - 5.4 | 8.11 (2.59) | 7.36 (2.64)
  DAS28 score >5.4 - 6.2 | 8.45 (2.19) | 7.58 (2.55)
  DAS28 score >6.2 | 8.31 (2.23) | 6.90 (2.85)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.749, Regression, Linear; Regression coefficient = 0.03, 95% CI 2-sided [-0.15 to 0.21]

14. Secondary Outcome: Participant Satisfaction by Participant's Global Assessment of RA Activity for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the delivery mechanism. Participants' global assessment of disease activity was measured on a visual analog scale (VAS) ranging from 0 (inactive) to 100 millimeter (mm) (extremely active). Results are reported by VAS scores observed for the participant's global assessment of RA activity: <=50 mm, >50-67 mm, >67-79 mm, >79 mm.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  VAS score for participant's assessment <=50 mm | 8.45 (2.14) | 7.55 (2.43)
  VAS score for participant's assessment >50 - 67 | 8.41 (2.15) | 7.31 (2.61)
  VAS score for participant's assessment >67 - 79 mm | 8.07 (2.60) | 7.11 (2.53)
  VAS score for participant's assessment >79 mm | 8.17 (2.59) | 6.88 (2.83)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.105, Regression, Linear; Regression coefficient = -0.08, 95% CI 2-sided [-0.18 to 0.02]

15. Secondary Outcome: Participant Satisfaction by Physician's Global Assessment of RA Activity for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. Physicians' global assessment of disease activity was measured on a VAS ranging from 0 (inactive) to 100 mm (extremely active). Results are reported by VAS scores observed for physician's global assessment of RA activity: <=47 mm, >47-61 mm, >61-72 mm, >72 mm.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  VAS score for physician's assessment <=47 mm | 8.23 (2.40) | 7.40 (2.24)
  VAS score for physician's assessment >47 - 61 mm | 8.36 (2.00) | 6.92 (2.73)
  VAS score for physician's assessment >61 - 72 mm | 8.03 (2.75) | 7.14 (2.96)
  VAS score for physician's assessment >72 mm | 8.47 (2.34) | 7.32 (2.59)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories; Test type: Superiority or Other; p = 0.819, Regression, Linear; Regression coefficient = 0.01, 95% CI 2-sided [-0.10 to 0.12]

16. Secondary Outcome: Participant Satisfaction by Health Assessment Questionnaire - Disability Index (HAQ-DI) for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. The 20-item HAQ-DI assessed the extent of participants' functional ability. Calculation yielded a single disability score from 0=normal or no difficulty to 3=unable to do. Lower HAQ-DI scores indicated better health. Results are reported by categories of HAQ-DI scores observed: <=0.9, >0.9-1.4, >1.4-1.9, >1.9.
Time Frame: Day 84
Population: mITT; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  HAQ-DI scale score <=0.9 | 8.61 (2.07) | 7.67 (2.24)
  HAQ-DI scale score >0.9 - 1.4 | 8.27 (2.37) | 7.40 (2.39)
  HAQ-DI scale score >1.4 - 1.9 | 8.33 (2.37) | 7.03 (2.84)
  HAQ-DI scale score >1.9 | 7.96 (2.58) | 6.57 (2.95)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; All categories, by 1-unit increments; Test type: Superiority or Other; p = 0.012, Regression, Linear; Regression coefficient = -0.39, 95% CI 2-sided [-0.69 to -0.09]

17. Secondary Outcome: Participant Satisfaction by Maximum Combination of Disease-Modifying Antirheumatic Drug (DMARD) Use for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the delivery mechanism. Participants were categorized into those who received only 1 DMARD, only 2 DMARDs, only 3 DMARDs, and at least 3 DMARDs.
Time Frame: Day 84
Population: mITT; LOCF. N=total evaluable participants. n=total evaluable participants for that category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 320 | 311
units on a scale
  1 DMARD (n=177, 162) | 8.29 (2.41) | 7.23 (2.66)
  2 DMARDs (n=123, 123) | 8.18 (2.42) | 7.19 (2.53)
  3 DMARDs (n=16, 26) | 8.94 (1.84) | 6.85 (3.04)
  At Least 4 DMARDs (n=4, 0) | 9.50 (1.00) | NA (NA) — NA=not available. This category had no participants, hence no data are available.
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; 2 DMARDs versus 1 DMARD (reference); Test type: Superiority or Other; p = 0.541, Regression, Linear; Regression coefficient = -0.10, 95% CI 2-sided [-0.52 to 0.32]
Statistical Analysis 2: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; 3 DMARDs versus 1 DMARD (reference); Test type: Superiority or Other; p = 0.541, Regression, Linear; Regression coefficient = -0.14, 95% CI 2-sided [-0.97 to 0.68]
Statistical Analysis 3: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; At least 4 DMARDs versus 1 DMARD (reference); Test type: Superiority or Other; p = 0.541, Regression, Linear; Regression coefficient = 1.72, 95% CI 2-sided [-0.82 to 4.25]

18. Secondary Outcome: Participant Satisfaction by Prior Injection Experience for 2 Different Delivery Mechanisms for Etanercept
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Participants were grouped into 2 categories: those who did and did not have prior injection experience. Higher scores indicated greater satisfaction with the delivery mechanism.
Time Frame: Day 84
Population: mITT; LOCF. n=evaluable participants in that category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 324 | 313
units on a scale
  Prior Injection Experience (n=177, 174) | 8.29 (2.35) | 7.05 (2.53)
  No Prior Injection Experience (n=147, 139) | 8.24 (2.42) | 7.37 (2.75)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Prior Injection Experience versus No Prior Injection Experience (reference); Test type: Superiority or Other; p = 0.465, Regression, Linear; Regression coefficient = -0.15, 95% CI 2-sided [-0.55 to 0.25]

19. Secondary Outcome: Short Form of the State-Trait Anxiety Inventory (SF-STAI) Global Score
Description: The SF-STAI consisted of 6 questions, each scored from 1 to 4. Total score ranged from 6=less anxiety to 24=more anxiety. Higher score indicated that the participant was more anxious.
Time Frame: Day 84
Population: mITT. N=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 303 | 298
units on a scale | 10.0 (3.7) | 10.5 (3.4)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.154, ANOVA; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.97 to 0.15], Standard Error of Mean 0.29

20. Secondary Outcome: Device Attributes and Participant Perception Questionnaire: How Satisfied Is the Subject With His/Her Life as a Whole?
Description: Score indicated satisfaction in response to the question "Thinking about your own life and personal circumstances, how satisfied are you with your life as a whole?" Score ranged from 0=completely dissatisfied to 10=completely satisfied. Higher scores indicated greater satisfaction.
Time Frame: Day 84
Population: mITT. N=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 307 | 300
units on a scale | 7.3 (2.2) | 7.1 (2.1)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.212, ANOVA; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.12 to 0.56], Standard Error of Mean 0.17

21. Secondary Outcome: Device Attributes and Participant Perception Questionnaire: How Satisfied Is the Subject With His/Her Health?
Description: Score indicated satisfaction in response to the question "How satisfied are you with your health?" Score ranged from 0=completely dissatisfied to 10=completely satisfied. Higher scores indicated greater satisfaction.
Time Frame: Day 84
Population: mITT. N=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 307 | 301
units on a scale | 6.1 (2.5) | 6.1 (2.4)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.965, ANOVA; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.39 to 0.37], Standard Error of Mean 0.19

22. Secondary Outcome: Device Attributes and Participant Perception Questionnaire: How Satisfied Is the Subject With All the Treatments He/She is Currently Receiving for RA?
Description: Score indicated satisfaction in response to the question "How satisfied are you with all the treatments you are currently receiving for your rheumatoid arthritis?" Score ranged from 0=completely dissatisfied to 10=completely satisfied. Higher scores indicated greater satisfaction.
Time Frame: Day 84
Population: mITT. N=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 307 | 301
units on a scale | 7.4 (2.4) | 7.3 (2.4)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.519, ANOVA; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.25 to 0.50], Standard Error of Mean 0.19

23. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 1, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Easy You Find the Device Is to Use - Q1: Overall, How Easy Was It to Perform an Injection with this Device? Participants specified their responses on a 5-point Likert scale: 0=very easy to 4=very difficult.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 298 | 295
percentage of participants
  0=Very Easy | 69.5 | 54.2
  1=Easy | 17.1 | 26.1
  2=Neither Easy nor Difficult | 7.0 | 12.5
  3=Difficult | 4.7 | 5.4
  4=Very Difficult | 1.7 | 1.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Day 84; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.33 to 2.57]

24. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 2, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Easy You Find the Device Is to Use - Q2: How Easy Was It to Learn to Use the Device? Participants specified their responses on a 5-point Likert scale: 0=very easy to 4=very difficult.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 295 | 294
percentage of participants
  0=Very Easy | 75.3 | 62.9
  1=Easy | 15.9 | 30.6
  2=Neither Easy nor Difficult | 5.4 | 5.1
  3=Difficult | 1.7 | 1.0
  4=Very Difficult | 1.7 | 0.3
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.007, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.14 to 2.29]

25. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 3, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Easy You Find the Device Is to Use - Q3: How Easy Is It to Dispose Of the Device? Participants specified their responses on a 5-point Likert scale: 0=very easy to 4=very difficult.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 288 | 291
percentage of participants
  0=Very Easy | 85.4 | 74.9
  1=Easy | 10.4 | 19.2
  2=Neither Easy nor Difficult | 2.4 | 4.8
  3=Difficult | 1.0 | 1.0
  4=Very Difficult | 0.7 | 0.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.002, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.26 to 2.92]

26. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 4, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Easy You Find the Device Is to Use - Q4: How Easy Is It to Know When the Injection Is Completed? Participants specified their responses on a 5-point Likert scale: 0=very easy to 4=very difficult.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 297 | 295
percentage of participants
  0=Very Easy | 81.1 | 63.4
  1=Easy | 13.1 | 26.1
  2=Neither Easy nor Difficult | 2.7 | 7.8
  3=Difficult | 2.7 | 2.4
  4=Very Difficult | 0.3 | 0.3
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.65 to 3.46]

27. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 5, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Easy You Find the Device Is to Use - Q5: How Easy Is It to Hold the Device Whilst Injecting? Participants specified their responses on a 5-point Likert scale: 0=very easy to 4=very difficult.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 292 | 294
percentage of participants
  0=Very Easy | 63.7 | 47.3
  1=Easy | 23.3 | 26.9
  2=Neither Easy nor Difficult | 7.9 | 16.0
  3=Difficult | 2.7 | 7.1
  4=Very Difficult | 2.4 | 2.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.50 to 2.83]

28. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 6, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Easy You Find the Device Is to Use - Q6: Did You Feel any Hand Discomfort Whilst Using the Device? Participants specified their responses on a 5-point Likert scale: 0=very easy to 4=very difficult.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 297 | 291
percentage of participants
  0=Very Easy | 69.0 | 54.3
  1=Easy | 18.5 | 19.9
  2=Neither Easy nor Difficult | 7.7 | 15.1
  3=Difficult | 3.4 | 7.6
  4=Very Difficult | 1.3 | 3.1
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.44 to 2.78]

29. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 7, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Easy You Find the Device Is to Use - Q7: How Long Does It Take to Perform the Injection, Including any Preparation and Disposal? Participants specified their responses on a 5-point Likert scale: 0=<5 minutes to 4=>30 minutes.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 295 | 295
percentage of participants
  <5 minutes | 64.7 | 57.6
  5-10 minutes | 22.0 | 30.8
  11-20 minutes | 6.8 | 6.8
  21-30 minutes | 5.1 | 3.7
  >30 minutes | 1.4 | 1.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.184, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.90 to 1.72]

30. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 8, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Convenient You Find the Device Is to Use - Q8: How Much Do You Think Injecting Etanercept Will Interfere with Your Ability to Enjoy Social or Leisure Activities? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 300
percentage of participants
  0=Not at all | 71.1 | 64.3
  1=A little | 14.3 | 17.7
  2=Somewhat | 7.0 | 11.3
  3=A lot | 4.7 | 4.7
  4=Very much | 3.0 | 2.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.106, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.94 to 1.85]

31. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 9, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Convenient You Find the Device Is to Use - Q9: Do You Think Injecting Etanercept Will Interfere with Your Usual Daily Activities? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 299
percentage of participants
  0=Not at all | 78.8 | 73.2
  1=A little | 12.3 | 15.7
  2=Somewhat | 5.6 | 5.7
  3=A lot | 2.3 | 4.3
  4=Very much | 1.0 | 1.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.112, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.93 to 1.96]

32. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 10, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Convenient You Find the Device Is to Use - Q10: How Much Do You Think Injecting Etanercept Will Interfere with Travelling on Holiday/ Business/Visiting? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 300
percentage of participants
  0=Not at all | 60.5 | 48.0
  1=A little | 20.6 | 23.0
  2=Somewhat | 9.3 | 17.7
  3=A lot | 7.0 | 7.7
  4=Very much | 2.7 | 3.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.002, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.21 to 2.24]

33. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 11, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Confident You Feel When Using the Device - Q11: Overall, How Confident Are You in Your Management of Your Weekly Injections? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 305 | 299
percentage of participants
  0=Not at all | 2.3 | 2.0
  1=A little | 1.6 | 5.4
  2=Somewhat | 6.2 | 8.4
  3=A lot | 22.0 | 30.4
  4=Very much | 67.9 | 53.8
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.41 to 0.78]

34. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 12, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Confident You Feel When Using the Device - Q12: How Confident Are You That You Inject the Right Amount of Medicine Every Time? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 305 | 300
percentage of participants
  0=Not at all | 1.3 | 1.3
  1=A little | 2.3 | 5.0
  2=Somewhat | 5.6 | 7.3
  3=A lot | 17.7 | 21.3
  4=Very much | 73.1 | 65.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.022, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.47 to 0.94]

35. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 13, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Confident You Feel When Using the Device - Q13: How Confident Are You That You Can Inject Yourself Properly with the Device? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 303 | 299
percentage of participants
  0=Not at all | 3.0 | 1.7
  1=A little | 3.0 | 6.0
  2=Somewhat | 5.9 | 8.4
  3=A lot | 17.2 | 23.4
  4=Very much | 71.0 | 60.5
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.009, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.46 to 0.89]

36. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 14, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Confident You Feel When Using the Device - Q14: Are You Confident That You Have Good Control over the Injection Process? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 305 | 299
percentage of participants
  0=Not at all | 2.3 | 1.7
  1=A little | 2.6 | 4.0
  2=Somewhat | 5.6 | 7.7
  3=A lot | 17.0 | 25.1
  4=Very much | 72.5 | 61.5
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.007, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.45 to 0.88]

37. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 15, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Confident You Feel When Using the Device - Q15: How Confident Are You That You Injected Yourself Successfully? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 304 | 299
percentage of participants
  0=Not at all | 2.6 | 1.0
  1=A little | 2.0 | 3.7
  2=Somewhat | 4.9 | 8.7
  3=A lot | 20.1 | 25.8
  4=Very much | 70.4 | 60.9
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.014, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.47 to 0.92]

38. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 16, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How You Feel When Using the Device - Q16: Overall, How Nervous Do You Feel about Your Injections? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 306 | 300
percentage of participants
  0=Not at all | 66.7 | 49.0
  1=A little | 19.3 | 25.3
  2=Somewhat | 8.8 | 15.0
  3=A lot | 3.6 | 7.0
  4=Very much | 1.6 | 3.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.53 to 2.88]

39. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 17, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How You Feel When Using the Device - Q17: Overall, How Nervous Do You Feel about Inserting the Needle into Your Skin? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 305 | 299
percentage of participants
  0=Not at all | 64.3 | 45.8
  1=A little | 21.3 | 27.8
  2=Somewhat | 6.9 | 12.4
  3=A lot | 5.9 | 8.4
  4=Very much | 1.6 | 5.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.57 to 2.91]

40. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 18, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How You Feel When Using the Device - Q18: Do You Dislike Injecting Yourself with this Device? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 305 | 300
percentage of participants
  0=Not at all | 70.8 | 46.0
  1=A little | 17.4 | 22.0
  2=Somewhat | 6.6 | 14.3
  3=A lot | 3.9 | 9.7
  4=Very much | 1.3 | 8.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 3.08, 95% CI 2-sided [2.23 to 4.25]

41. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 19, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How You Feel When Using the Device - Q19: Overall, Are You Emotionally Distressed or Anxious about Your Injections? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 306 | 299
percentage of participants
  0=Not at all | 70.6 | 57.2
  1=A little | 18.0 | 22.7
  2=Somewhat | 7.2 | 8.7
  3=A lot | 2.3 | 6.4
  4=Very much | 2.0 | 5.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.35 to 2.62]

42. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 20, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: What Characteristics of the Device You Appreciate - Q20: How Much Do You Like the Look of the Device? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 304 | 298
percentage of participants
  0=Not at all | 1.6 | 10.4
  1=A little | 3.6 | 10.1
  2=Somewhat | 19.4 | 35.9
  3=A lot | 32.6 | 24.8
  4=Very much | 42.8 | 18.8
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.18 to 0.34]

43. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 21, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: What Characteristics of the Device You Appreciate - Q21: How Much Do You Like the Feel of the Device? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 304 | 296
percentage of participants
  0=Not at all | 3.0 | 9.5
  1=A little | 3.0 | 10.8
  2=Somewhat | 20.1 | 35.1
  3=A lot | 33.6 | 27.0
  4=Very much | 40.5 | 17.6
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.19 to 0.36]

44. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 22, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: What Characteristics of the Device You Appreciate - Q22: How Much Does the Device Look Like Something You Would Feel Comfortable to Use? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 297
percentage of participants
  0=Not at all | 4.0 | 12.1
  1=A little | 3.6 | 8.8
  2=Somewhat | 18.2 | 31.6
  3=A lot | 27.5 | 29.0
  4=Very much | 46.7 | 18.5
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.20 to 0.36]

45. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 23, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: Side Effects from Using the Device - Q23: Do You Experience Pain During or Immediately After the Injection? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 304 | 298
percentage of participants
  0=Not at all | 36.2 | 39.6
  1=A little | 28.0 | 29.9
  2=Somewhat | 20.4 | 17.8
  3=A lot | 11.8 | 9.1
  4=Very much | 3.6 | 3.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.196, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.61 to 1.11]

46. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 24, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Likely Is It That You Would Use the Device Again - Q24: To What Extent Would You Consider Alternative Devices If You Were to Continue on Etanercept? Participants specified their responses on a 5-point Likert scale: 0=very little to 4=very much.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 240 | 232
percentage of participants
  0=Very little | 48.8 | 28.4
  1=A little | 8.8 | 21.1
  2=Somewhat | 20.8 | 22.8
  3=A lot | 8.3 | 11.2
  4=Very much | 13.3 | 16.4
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p = 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.25 to 2.42]

47. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 25, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Likely Is It That You Would Use the Device Again - Q25: Would You Recommend this Device to Someone Else Who Needed to Self Inject? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=yes definitely.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 296
percentage of participants
  0=Not at all | 3.3 | 4.4
  1=Rarely | 2.3 | 5.4
  2=Occasionally | 7.6 | 24.7
  3=Often | 12.3 | 19.3
  4=Yes definitely | 74.4 | 46.3
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.21 to 0.42]

48. Secondary Outcome: Percentage of Participants Responding to the Device Attribute and Participant Questionnaire, Question 26, Day 84
Description: Percentage of participants responding to Device Attributes and Subject Perceptions Questionnaire: How Likely Is It That You Would Use the Device Again - Q26: If Your Doctor Advised You to, How Likely Would You to Be Continue Injecting Regularly With this Device? Participants specified their responses on a 5-point Likert scale: 0=not at all to 4=very likely.
Time Frame: Day 84
Population: mITT. N=participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 297
percentage of participants
  0=Not at all | 3.0 | 3.7
  1=Usually not | 3.0 | 7.7
  2=Occasionally | 9.3 | 17.8
  3=Likely | 11.0 | 18.9
  4=Very likely | 73.8 | 51.9
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector vs Enbrel 50 mg Prefilled Syringe; Test type: Superiority or Other; p < 0.001, GEE model+logit link+multinomial distrib; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.29 to 0.56]

49. Secondary Outcome: Age Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The mean age was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 age clusters who reported themselves as being very satisfied, satisfied, or not satisfied. n=number of participants who reported themselves as being very satisfied, satisfied, or not satisfied for the specified treatment arm.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 296
years
  Cluster 1, Very Satisfied (n=204, 133) | 54.3 (12.3) | 56.0 (13.0)
  Cluster 2, Satisfied (n=51, 71) | 55.1 (11.9) | 54.1 (12.5)
  Cluster 3, Not Satisfied (n=47, 92) | 54.0 (14.6) | 52.7 (13.2)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.896, ANOVA
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.166, ANOVA

50. Secondary Outcome: Percentage of Male Participants Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, all male and female participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The percentage of participants who were male was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. n=number of participants (male plus female) who reported themselves as being very satisfied, satisfied, or not for the specified treatment arm.
Measure: Number; unit: percentage of male participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 296
percentage of male participants
  Cluster 1, Very Satisfied (n=204, 133) | 30.9 | 30.1
  Cluster 2, Satisfied (n=51, 71) | 23.5 | 29.6
  Cluster 3, Not Satisfied (n=47, 92) | 14.9 | 14.1
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.069, Chi-squared
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.015, Chi-squared

51. Secondary Outcome: Percentage of Female Participants Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, all male and female participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Percentage of participants who were female was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants (male+female) across all 3 clusters who reported themselves as being very satisfied, satisfied, or not satisfied. n=number of participants (male+female) who reported themselves as being very satisfied, satisfied, or not satisfied for the specified treatment arm and gender.
Measure: Number; unit: percentage of female participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 296
percentage of female participants
  Cluster 1, Very Satisfied (n=204, 133) | 69.1 | 69.9
  Cluster 2, Satisfied (n=51, 71) | 76.5 | 70.4
  Cluster 3, Not Satisfied (n=47, 92) | 85.1 | 85.9
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.069, Chi-squared
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.015, Chi-squared

52. Secondary Outcome: Percentage of Participants With Only Reading/Writing Capacity Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants in all 3 social-educational level (only reading/writing capacity, high-school level, university level) were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Percentage of participants with only reading/writing capacity was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 social-educational levels and across all 3 clusters who reported themselves as very satisfied, satisfied, or not satisfied. n=participants across all 3 levels reporting themselves as very satisfied, satisfied, or not satisfied for the specified treatment arm.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 294
percentage of participants
  Cluster 1, Very Satisfied (n=203, 132) | 35.0 | 44.7
  Cluster 2, Satisfied (n=51, 70) | 45.1 | 42.9
  Cluster 3, Not Satisfied (n=47, 92) | 36.2 | 33.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.652, Chi-squared
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.459, Chi-squared

53. Secondary Outcome: Percentage of Participants at High School/Baccalaureate Level Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants in all 3 social-educational level (only reading/writing capacity, high-school level, university level) were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Percentage of participants at high school/baccalaureate level was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 social-educational levels and across all 3 clusters who reported themselves as very satisfied, satisfied, or not satisfied. n=participants at all 3 levels reporting themselves as very satisfied, satisfied, or not satisfied for the specified treatment arm.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 294
percentage of participants
  Cluster 1, Very Satisfied (n=203, 132) | 48.8 | 43.2
  Cluster 2, Satisfied (n=51, 70) | 37.3 | 41.4
  Cluster 3, Not Satisfied (n=47, 92) | 48.9 | 47.8
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.652, Chi-squared
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.459, Chi-squared

54. Secondary Outcome: Percentage of Participants at University Level Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants in all 3 social-educational level (only reading/writing capacity, high-school level, university level) were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Percentage of participants at the university level was determined for each cluster of participants.
Time Frame: Day 84
Population: as for outcome 52
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 294
percentage of participants
  Cluster 1, Very Satisfied (n=203, 132) | 16.3 | 12.1
  Cluster 2, Satisfied (n=51, 70) | 17.6 | 15.7
  Cluster 3, Not Satisfied (n=47, 92) | 14.9 | 18.5
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.652, Chi-squared
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.459, Chi-squared

55. Secondary Outcome: HAD Anxiety Subscale Score Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The mean HAD Anxiety Subscale Score was determined for each cluster of participants. Score ranged from 0 to 21. Lower scores indicated better health.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 clusters who reported themselves as being very satisfied, satisfied, or not satisfied. n=number of participants who reported themselves as being very satisfied, satisfied, or not satisfied for the specified treatment arm and cluster.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 295
units on a scale
  Cluster 1, Very Satisfied (n=203, 132) | 6.8 (4.2) | 6.4 (4.5)
  Cluster 2, Satisfied (n=51, 71) | 7.9 (3.8) | 7.4 (4.0)
  Cluster 3, Not Satisfied (n=47, 92) | 8.3 (3.7) | 8.7 (3.8)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.023, Kruskal-Wallis
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

56. Secondary Outcome: HAD Depression Subscale Score Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The mean HAD Depression Subscale Score was determined for each cluster of participants. Score ranged from 0 to 21. Lower scores indicated better health.
Time Frame: Day 84
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 301 | 296
units on a scale
  Cluster 1, Very Satisfied (n=203, 133) | 5.8 (3.8) | 5.0 (3.9)
  Cluster 2, Satisfied (n=51, 71) | 6.6 (3.9) | 5.2 (3.5)
  Cluster 3, Not Satisfied (n=47, 92) | 7.3 (4.1) | 6.7 (3.6)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.038, Kruskal-Wallis
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

57. Secondary Outcome: PAM Score Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The mean PAM Score was determined for each cluster of participants. Calibrated PAM scale score ranged from 0 to 100.Higher scores indicated more confidence in managing participants' condition and lifestyle.
Time Frame: Day 84
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 296 | 293
units on a scale
  Cluster 1, Very Satisfied (n=198, 131) | 61.6 (13.1) | 60.1 (14.0)
  Cluster 2, Satisfied (n=51, 71) | 56.6 (11.5) | 56.5 (11.7)
  Cluster 3, Not Satisfied (n=47, 91) | 57.4 (13.8) | 55.3 (11.9)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.018, ANOVA
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.019, ANOVA

58. Secondary Outcome: Percentage of Participants With Prior Injection Experience Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The percentage of participants with prior injection experience was determined for each cluster of participants.
Time Frame: Day 84
Population: as for outcome 55
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 296
percentage of participants
  Cluster 1, Very Satisfied (n=204, 133) | 52.9 | 54.9
  Cluster 2, Satisfied (n=51, 71) | 47.1 | 54.9
  Cluster 3, Not Satisfied (n=47, 92) | 70.2 | 59.8
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.049, Chi-squared
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.736, Chi-squared

59. Secondary Outcome: Percentage of Participants With Prior Self-Injection Experience Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. The percentage of participants with prior self-injection experience was determined for each cluster of participants.
Time Frame: Day 84
Population: as for outcome 55
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 296
percentage of participants
  Cluster 1, Very Satisfied (n=204, 133) | 31.9 | 31.6
  Cluster 2, Satisfied (n=51, 71) | 15.7 | 36.6
  Cluster 3, Not Satisfied (n=47, 92) | 38.3 | 31.5
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.033, Chi-squared
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.730, Chi-squared

60. Secondary Outcome: RA Duration Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The mean RA Duration was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 clusters who reported themselves as being very satisfied, satisfied, or not satisfied. n=number of participants who reported themselves as being very satisfied, satisfied , or not satisfied for the specified treatment arm and cluster.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 296
years
  Cluster 1, Very Satisfied (n=204, 133) | 8.6 (8.0) | 9.7 (9.1)
  Cluster 2, Satisfied (n=51, 71) | 9.4 (8.2) | 8.6 (8.1)
  Cluster 3, Not Satisfied (n=47, 92) | 8.9 (8.9) | 10.3 (8.4)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.838, ANOVA
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.483, ANOVA

61. Secondary Outcome: DAS28 Score Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The mean DAS28 Score was determined for each cluster of participants. Score ranged from 0 to 9.4. Interpretation: disease activity is low when score ≤3.2, moderate when 3.2<score≤5.1, or high when score >5.1, remission when score <2.6.
Time Frame: Day 84
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 292 | 287
units on a scale
  Cluster 1, Very Satisfied (n=197, 128) | 5.3 (1.1) | 5.5 (1.1)
  Cluster 2, Satisfied (n=50, 70) | 5.4 (1.3) | 5.0 (1.3)
  Cluster 3, Not Satisfied (n=45, 89) | 5.5 (1.1) | 5.5 (1.2)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.466, Kruskal-Wallis
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.035, Kruskal-Wallis

62. Secondary Outcome: Participant's Global Assessment of RA Activity Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Participants' mean Global Assessment of RA Activity was determined for each cluster of participants. VAS scores ranged from 0 (inactive) to 100 mm (extremely active).
Time Frame: Day 84
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: millimeters on the VAS
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 298 | 294
millimeters on the VAS
  Cluster 1, Very Satisfied (n=202, 132) | 63.5 (20.2) | 62.5 (21.4)
  Cluster 2, Satisfied (n=50, 71) | 64.7 (19.2) | 57.5 (24.0)
  Cluster 3, Not Satisfied (n=46, 91) | 65.7 (19.5) | 68.2 (17.6)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.784, ANOVA
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.006, ANOVA

63. Secondary Outcome: Physician's Global Assessment of RA Activity Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Mean Physician's Global Assessment of RA Activity was determined for each cluster of participants. VAS scores ranged from 0 (inactive) to 100 mm (extremely active).
Time Frame: Day 84
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: millimeters on the VAS
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 299 | 295
millimeters on the VAS
  Cluster 1, Very Satisfied (n=203, 132) | 58.8 (18.6) | 60.8 (19.0)
  Cluster 2, Satisfied (n=50, 71) | 58.3 (18.3) | 57.4 (21.6)
  Cluster 3, Not Satisfied (n=46, 92) | 60.3 (16.8) | 60.1 (16.6)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.843, ANOVA
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.461, ANOVA

64. Secondary Outcome: HAQ-DI Score Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. The mean HAQ-DI Score, assessing the extent of functional ability, was determined for each cluster of participants. Disability score ranged from 0=normal or no difficulty to 3=unable to do. Lower HAQ-DI scores indicated better health.
Time Frame: Day 84
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 300 | 296
units on a scale
  Cluster 1, Very Satisfied (n=204, 133) | 1.4 (0.7) | 1.3 (0.7)
  Cluster 2, Satisfied (n=51, 71) | 1.5 (0.6) | 1.3 (0.6)
  Cluster 3, Not Satisfied (n=45, 92) | 1.5 (0.6) | 1.6 (0.6)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.150, Kruskal-Wallis
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.002, Kruskal-Wallis

65. Secondary Outcome: Percentage of Participants Receiving Only 1 DMARD Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, all participants receiving DMARDs (only 1, only 2, only 3, 4 or more DMARDs) were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Percentage of participants receiving only 1 DMARD was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 clusters receiving only 1 DMARD who reported themselves as being very satisfied, satisfied, or not satisfied. n=number of participants who reported themselves as being very satisfied, satisfied , or not satisfied for the specified treatment arm and cluster.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 163 | 155
percentage of participants
  Cluster 1, Very Satisfied (n=112, 73) | 55.4 | 55.3
  Cluster 2, Satisfied (n=26, 38) | 52.0 | 53.5
  Cluster 3, Not Satisfied (n=25, 44) | 54.3 | 48.4
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.934, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.656, Cochran-Mantel-Haenszel

66. Secondary Outcome: Percentage of Participants Receiving Only 2 DMARDs Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, all participants receiving DMARDs (only 1, only 2, only 3, 4 or more DMARDs) were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Percentage of participants receiving only 2 DMARDs was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 clusters receiving only 2 DMARDs, who reported themselves as very satisfied, satisfied, or not satisfied. n=number of participants receiving only 2 DMARDs who reported themselves as being very satisfied, satisfied , or not satisfied for the specified treatment arm.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 117 | 115
percentage of participants
  Cluster 1, Very Satisfied (n=77, 49) | 38.1 | 37.1
  Cluster 2, Satisfied (n=21, 26) | 42.0 | 36.6
  Cluster 3, Not Satisfied (n=19, 40) | 41.3 | 44.0
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.934, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.656, Cochran-Mantel-Haenszel

67. Secondary Outcome: Percentage of Participants Receiving Only 3 DMARDs Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, all participants receiving DMARDs (only 1, only 2, only 3, 4 or more DMARDs) were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Percentage of participants receiving only 3 DMARDs was determined for each cluster of participants.
Time Frame: Day 84
Population: mITT. Number of participants analyzed (N)=total number of participants across all 3 clusters receiving only 3 DMARDs who reported themselves as being very satisfied, satisfied, or not satisfied. n=number of participants receiving only 3 DMARDs who reported themselves as very satisfied, satisfied , or not satisfied for the specified treatment arm.
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 14 | 24
percentage of participants
  Cluster 1, Very Satisfied (n=9, 10) | 4.5 | 7.6
  Cluster 2, Satisfied (n=3, 7) | 6.0 | 9.9
  Cluster 3, Not Satisfied (n=2, 7) | 4.3 | 7.7
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p = 0.934, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p = 0.656, Cochran-Mantel-Haenszel

68. Secondary Outcome: Participant Satisfaction at Endpoint Associated With Participant Perception
Description: Participant perception was assessed with the 26 questions in the Device Attribute and Participant Questionnaire. Based on the scores assigned to the 26 questions, participants were grouped into 3 clusters (Cluster 1=very satisfied, Cluster 2=satisfied, Cluster 3=not satisfied) using multiple correspondence analysis and ascending hierarchical classification. Mean participant satisfaction was determined for each cluster of participants. Satisfaction was scored on a 10-point scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction.
Time Frame: Day 84
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Number analyzed (Participants) | 302 | 296
units on a scale
  Cluster 1, Very Satisfied (n=204, 133) | 9.0 (1.9) | 8.0 (2.5)
  Cluster 2, Satisfied (n=51, 71) | 8.1 (1.7) | 8.2 (1.6)
  Cluster 3, Not Satisfied (n=47, 92) | 5.5 (2.8) | 5.3 (2.4)
Statistical Analysis 1: Comparison: Enbrel 50 mg Autoinjector; p-value for statistical difference between 3 clusters in the Autoinjector group; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Enbrel 50 mg Prefilled Syringe; p-value for statistical difference between 3 clusters in the Prefilled Syringe group; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Enbrel 50 mg Autoinjector | Enbrel 50 mg Prefilled Syringe
Serious Adverse Events (participants affected / at risk) | 18/325 | 9/313
Other Adverse Events (participants affected / at risk) | 203/325 | 201/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enbrel 50 mg Autoinjector (N=325) | Enbrel 50 mg Prefilled Syringe (N=313)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Complication of device insertion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cervical root pain (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Breast cyst excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enbrel 50 mg Autoinjector (N=325) | Enbrel 50 mg Prefilled Syringe (N=313)
Nausea (Gastrointestinal disorders) | 7 (8) | 9 (32)
Injection site erythema (General disorders) | 25 (61) | 29 (62)
Injection site haematoma (General disorders) | 15 (19) | 6 (6)
Injection site haemorrhage (General disorders) | 10 (14) | 6 (6)
Injection site irritation (General disorders) | 3 (3) | 10 (20)
Injection site pain (General disorders) | 20 (43) | 13 (30)
Injection site rash (General disorders) | 3 (6) | 7 (9)
Injection site reaction (General disorders) | 46 (97) | 55 (173)
Bronchitis (Infections and infestations) | 6 (7) | 12 (13)
Influenza (Infections and infestations) | 9 (9) | 8 (8)
Nasopharyngitis (Infections and infestations) | 22 (22) | 26 (28)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 9 (10)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (10)
Headache (Nervous system disorders) | 9 (15) | 6 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 9 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.